CLINICAL TRIAL: NCT06937476
Title: Investigation of the Neurobiological Mechanisms Underlying Pathological Rumination and the Pharmacological Effects of Aripiprazole
Brief Title: Neurobiological Mechanisms of Pathological Rumination and Effects of Aripiprazole
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Collaborators: Second Xiangya Hospital of Central South University (Other); National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Zhang Yan, Principal Investigator, Department of Psychiatry, The Second Xiangya Hospital, Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LYG20230074
Record Dates: First submitted 2025-04-20; First posted 2025-04-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder (MDD); Rumination
Keywords: Aripiprazole; Neuroimaging; Dopaminergic pathway; Fallypride; Randomized Controlled Trial; Cognitive symptoms; D2 receptor; PET-MRI
MeSH Terms: conditions — Depressive Disorder, Major; Rumination Syndrome; Neurobehavioral Manifestations | interventions — Escitalopram; Aripiprazole

STUDY DESIGN:
Intervention Model Description: This study involves four parallel groups: (1) pathological-rumination MDD patients treated with escitalopram alone (n=24), (2) pathological-rumination MDD patients treated with escitalopram plus aripiprazole (n=24), (3) non-pathological-rumination MDD patients without intervention (n=24), and (4) healthy controls without intervention (n=36). The increased sample size of the healthy control group is intended to provide a representative normative reference for clinical and imaging measures.
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessors and data analysts will be blinded to treatment allocation. Study participants and clinical investigators will remain unblinded due to the need for dosage adjustment and monitoring. Rater blinding is maintained to reduce assessment bias in outcome measures such as the Ruminative Responses Scale (RRS) and Hamilton Depression Rating Scale (HAMD).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Escitalopram Only - MDD with Pathological Rumination (Experimental): Patients diagnosed with major depressive disorder (MDD) and exhibiting pathological rumination will receive escitalopram monotherapy at 20 mg/day for 8 weeks.
  Interventions: Drug: Escitalopram
- Escitalopram + Aripiprazole - MDD with Pathological Rumination (Experimental): Patients with MDD and pathological rumination will receive escitalopram (20 mg/day) and low-dose aripiprazole (2.5-5 mg/day) for 8 weeks, with titration based on tolerability.
  Interventions: Drug: Escitalopram; Drug: Aripiprazole 5mg
- MDD with Low Rumination - Observational (No Intervention): MDD patients with low levels of rumination (RRS < 61) will receive no pharmacological intervention and serve as a naturalistic observation group.
- Healthy Controls (No Intervention): Healthy individuals with no psychiatric history will serve as non-clinical imaging and behavioral controls.

INTERVENTIONS:
Drug: Escitalopram — Escitalopram will be administered orally at a fixed dose of 20 mg/day for 8 weeks. This SSRI antidepressant is used as baseline pharmacological treatment for patients with major depressive disorder (MDD), either as monotherapy or in combination with aripiprazole. No other psychotropic medications are allowed during the study period.
  Arms: Escitalopram + Aripiprazole - MDD with Pathological Rumination; Escitalopram Only - MDD with Pathological Rumination
Drug: Aripiprazole 5mg — Aripiprazole will be administered as an adjunctive treatment to escitalopram at an initial dose of 2.5 mg/day, titrated up to 5 mg/day based on tolerability. Treatment will last 8 weeks, after which aripiprazole will be tapered and discontinued. This intervention aims to evaluate the efficacy of dopaminergic augmentation in reducing pathological rumination symptoms.
  Arms: Escitalopram + Aripiprazole - MDD with Pathological Rumination

SUMMARY:
This randomized, single-blind (assessor-blind) controlled trial aims to investigate the efficacy of aripiprazole as an augmentation strategy for treating pathological rumination in patients with major depressive disorder (MDD). Pathological rumination-defined as repetitive, intrusive, and uncontrollable negative thinking-has been identified as a major transdiagnostic risk factor for the development, maintenance, and recurrence of depression. Even during clinical remission, ruminative symptoms often persist and strongly predict relapse.

Previous clinical observations and experimental studies suggest that aripiprazole, a partial dopamine D2 receptor agonist, can significantly improve cognitive symptoms and reduce rumination in MDD patients when added to selective serotonin reuptake inhibitors (SSRIs). However, rigorous randomized controlled trials (RCTs) directly targeting rumination and validating this effect remain limited.

In this study, patients with acute MDD episodes and high levels of rumination will be randomly assigned to receive either escitalopram monotherapy (20 mg/day) or escitalopram (20 mg/day) plus low-dose aripiprazole (2.5-5 mg/day) for 8 weeks. The assignment will remain blinded to outcome assessors and data analysts, while patients and treating clinicians will remain unblinded due to dose titration and safety monitoring requirements.

Participants will undergo [18F]fallypride-PET-MRI scanning at baseline and post-treatment to measure striatal dopamine D2 receptor binding and explore its association with changes in rumination symptoms and treatment efficacy.

The primary outcome is the change in Ruminative Responses Scale (RRS) scores. Secondary outcomes include changes in depressive symptoms and dopamine D2 receptor availability. This trial will provide neurobiological insights into the dopaminergic mechanisms underlying pathological rumination and explore the therapeutic potential of D2 receptor modulation in this cognitive domain.

DETAILED DESCRIPTION:
Revised Detailed Description（Single-Blind Assessor-Blind Version）

Background:

Pathological rumination is characterized by repetitive, intrusive, and difficult-to-control negative thinking that often persists even after depressive symptoms remit. It has been recognized as a proximal risk factor for the onset, maintenance, and recurrence of major depressive disorder (MDD). Recent meta-analyses and longitudinal studies have confirmed that rumination significantly contributes to poor treatment outcomes and is associated with trait-like persistence across diagnostic and symptomatic states.

Rationale:

Aripiprazole, a partial dopamine D2 receptor agonist, has shown potential in augmenting antidepressant therapy by improving cognitive control and reducing rumination. Clinical observations have suggested that adjunctive aripiprazole can significantly alleviate ruminative symptoms in MDD patients, yet high-quality randomized controlled trials (RCTs) directly targeting rumination as a primary outcome remain lacking. Dopaminergic dysfunction-particularly altered D2 receptor availability in the striatum-may underlie the neurobiological mechanisms of pathological rumination. Therefore, combining pharmacological intervention with molecular neuroimaging offers a promising translational approach to validate therapeutic targets.

Study Design:

This study adopts a randomized, single-blind (assessor-blind) controlled trial design. Eligible participants include unmedicated or drug-naive MDD patients with high levels of rumination and healthy controls. Patients with pathological rumination will be randomly assigned to one of two intervention arms:

Group I: Escitalopram (20 mg/day) + aripiprazole (2.5-5 mg/day) Group II: Escitalopram monotherapy (20 mg/day)

The aripiprazole dose will be titrated from 2.5 mg/day to a maximum of 5 mg/day based on tolerability. During weeks 9-10, aripiprazole will be tapered and discontinued, with escitalopram maintained. No additional psychotropic medications are allowed. Outcome assessors and data analysts will remain blinded to treatment allocation to minimize assessment bias.

Neuroimaging Assessment:

Participants will undergo two [18F]fallypride-PET-MRI scans (at baseline and at the end of treatment in week 8). The scanning protocol includes:

Intravenous injection of 5 mCi [18F]-fallypride Dynamic PET acquisition in three blocks (70 min, 50 min, 60 min) with resting intervals Image reconstruction of binding potential (BPND) maps using simplified reference tissue modeling (SRTM), with the cerebellum as the reference region

Outcome Measures:

Primary outcome: Change in Ruminative Responses Scale (RRS) score Secondary outcomes: Changes in depressive symptoms (e.g., HAMD), striatal D2 receptor BPND values, and the correlations between imaging changes and clinical improvement

Hypothesis:

Aberrant striatal dopamine D2 receptor availability is a neurobiological substrate of pathological rumination. Modulating D2 receptor activity via aripiprazole can reduce rumination and enhance treatment response. Neuroimaging markers are expected to correlate with symptom improvement, providing mechanistic insight into the dopaminergic contributions to depressive cognition.

ELIGIBILITY:
Inclusion Criteria:

* For Patients with Major Depressive Disorder (MDD):

Age 18 to 45 years old, any sex.

Han Chinese, right-handed.

Education level of junior high school or above, able to understand informed consent and complete self-report instruments.

Meets DSM-5 diagnostic criteria for Major Depressive Disorder (MDD) based on the SCID interview.

Currently experiencing a depressive episode:

HAMD-24 score ≥ 21

YMRS score ≤ 5

No psychotropic medication (except benzodiazepines) in the past 6 weeks.

Classified into one of two cognitive subgroups based on rumination:

Pathological Rumination Group: Must meet all three of the following:

1. Subjective experience (e.g., "I can't stop thinking about past regrets" or "I can't control painful thoughts...")
2. Interview-confirmed features of pathological rumination (all of the following):

   Repetitive Intrusive Difficult to disengage Unproductive Capturing mental capacity
3. Ruminative Responses Scale (RRS) score ≥ 61

Low Rumination Group: Does not meet the above criteria.

Exclusion Criteria:

* Meets DSM-5 criteria for psychiatric disorders other than anxiety disorders.

MDD with psychotic features.

Severe suicidal ideation or behavior.

History of traumatic brain injury or loss of consciousness.

Serious neurological or medical illness (e.g., thyroid disorders, lupus, diabetes, infection, trauma).

Cardiac pacemaker or any metallic implants incompatible with MRI/PET.

History of alcohol or substance dependence.

Pregnant or breastfeeding.

Personal or family history of epilepsy.

Underwent non-pharmacological psychiatric interventions (e.g., ECT, rTMS, psychotherapy) in the past 6 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Ruminative Responses Scale (RRS) score from baseline to week 8 | Baseline and week 8
  The Ruminative Responses Scale (RRS) will be used to assess the severity of pathological rumination. The primary outcome is the change in total RRS score from baseline to the end of the 8-week treatment period. Higher scores indicate more severe rumination.

SECONDARY OUTCOMES:
Change in 24-item Hamilton Depression Rating Scale (HAMD-24) score | Baseline and week 8
  Depression severity will be assessed using the 24-item HAMD. The outcome is the change in total score from baseline to week 8. This will help evaluate overall clinical improvement in depressive symptoms.

OTHER OUTCOMES:
Exploratory multimodal biomarkers (MRI, blood, urine, stool), neurocognition, and additional symptom questionnaires | Baseline and week 8
  MRI (T1, BOLD fMRI, diffusion NODDI, NM-MRI) will generate prespecified imaging-derived metrics for exploratory analyses. Blood will be assayed for selected inflammatory, neurotrophic, neuroendocrine, and metabolic biomarkers (e.g., hs-CRP, IL-6, TNF-α, BDNF, cortisol, fasting glucose, lipids) for exploratory biomarker analyses. Urine and stool will be collected for exploratory biomarkers/omics, including urine metabolomic metrics and gut microbiome measures (e.g., diversity indices and taxonomic relative abundance; optional short-chain fatty acids [SCFAs]). Neurocognition will be evaluated with a standardized test battery (composite and/or domain scores). Questionnaires include HAMA, HAMD-24, MADRS, BSI, YMRS, Depression Symptom Rapid Self-rating, GAD-7, PHQ-9, PSQI, CTQ, STAI, Perceived Stress Scale, PCL-5, CERQ, DERS, RRS, PTQ, PSWQ, BSRI, DAS, Resilience Scale, PDQ-D, Treatment Adherence Scale, and SHAPS.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the published results (including de-identified clinical and imaging data) will be available upon reasonable request from qualified researchers. Data will be shared after publication, with prior approval from the corresponding author and ethical oversight. Supporting documents such as the study protocol and statistical analysis plan will also be made available where applicable.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data (IPD) and supporting documents will be available beginning 6 months after publication of the main results and will remain available for up to 5 years, or as long as the dataset is maintained by the research team.
Access Criteria: De-identified clinical and imaging data will be made available to qualified researchers with a methodologically sound proposal, subject to approval by the principal investigator and institutional ethics board. Data requests can be submitted by email and will require signing a data use agreement.

REFERENCES:
- [Background] van der Velden AM, Scholl J, Elmholdt EM, Fjorback LO, Harmer CJ, Lazar SW, O'Toole MS, Smallwood J, Roepstorff A, Kuyken W. Mindfulness Training Changes Brain Dynamics During Depressive Rumination: A Randomized Controlled Trial. Biol Psychiatry. 2023 Feb 1;93(3):233-242. doi: 10.1016/j.biopsych.2022.06.038. Epub 2022 Jul 22. PMID 36328822
- [Background] Song AK, Hay KR, Trujillo P, Aumann M, Stark AJ, Yan Y, Kang H, Donahue MJ, Zald DH, Claassen DO. Amphetamine-induced dopamine release and impulsivity in Parkinson's disease. Brain. 2022 Oct 21;145(10):3488-3499. doi: 10.1093/brain/awab487. PMID 34951464
- [Background] Wang Y, Lu Z, Xun G. Effect of aripiprazole on promoting cognitive function and enhancing clinical efficacy in patients with first-episode depression on escitalopram: A randomized controlled trial. J Affect Disord. 2024 Jan 1;344:159-168. doi: 10.1016/j.jad.2023.10.038. Epub 2023 Oct 10. PMID 37827257
- [Background] Ehring T. Thinking too much: rumination and psychopathology. World Psychiatry. 2021 Oct;20(3):441-442. doi: 10.1002/wps.20910. No abstract available. PMID 34505392